CLINICAL TRIAL: NCT00633984
Title: D-Cycloserine Enhancement of Exposure in Social Phobia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Boston University (Other); Southern Methodist University (Other); National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Mark H. Pollack, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2007-P-000386; R01MH075889 (NIH)
Record Dates: First submitted 2008-03-04; First posted 2008-03-12 (Estimated); Results first posted 2014-05-14 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-04

CONDITIONS: Social Anxiety Disorder
Keywords: Social Anxiety Disorder; Cognitive Behavioral Group Therapy; D-cycloserine
MeSH Terms: conditions — Phobia, Social | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Behavioral Group Therapy + D-Cycloserine (Active Comparator): Participants received Cognitive Behavioral Group Therapy and 50mg D-Cycloserine.
  Interventions: Behavioral: Cognitive Behavioral Group Therapy (CBGT); Drug: D-Cycloserine
- Cognitive Behavioral Group Therapy + Placebo (Placebo Comparator): Participants received Cognitive Behavioral Group Therapy and 50mg Placebo.
  Interventions: Behavioral: Cognitive Behavioral Group Therapy (CBGT); Drug: Placebo

INTERVENTIONS:
Behavioral: Cognitive Behavioral Group Therapy (CBGT) — The patient will then receive 12 weekly sessions of Cognitive Behavioral Therapy lasting approximately two and a half hours each. During these sessions, patients will receive information on the nature of social phobia and a model of treatment and will receive weekly training in how to become more comfortable with social situations, with the goal of achieving confidence in social interactions. As part of this training, the therapist will practice social interactions with the patient, who will also be asked to practice what they have learned outside of the therapists' office.
Drug: D-Cycloserine — For the third, fourth, fifth, sixth, and seventh sessions of the twelve-session program of Cognitive Behavioral Therapy, the patient will be asked to arrive one hour early to take one of the study pill, a 50mg pill of d-cycloserine. A physician will be available in the unlikely event that a patient begins to experience side effects. Before the treatment starts, before the eighth session, and one week after the final session patients will have a separate visit in which their levels of symptoms assessed with measures of mood, anxiety, and avoidance.
  Arms: Cognitive Behavioral Group Therapy + D-Cycloserine
Drug: Placebo — For the third, fourth, fifth, sixth, and seventh sessions of the twelve-session program of Cognitive Behavioral Therapy, the patient will be asked to arrive one hour early to take one of the study pill, a placebo. A physician will be available in the unlikely event that a patient begins to experience side effects. Before the treatment starts, before the eighth session, and one week after the final session patients will have a separate visit in which their levels of symptoms assessed with measures of mood, anxiety, and avoidance.
  Arms: Cognitive Behavioral Group Therapy + Placebo

SUMMARY:
The purpose of this study is to test a drug called d-cycloserine to see if it can help people with a condition called social phobia. Social phobia is also called "social anxiety disorder." Social phobia is a constant fear of social or performance situations. Social situations include group gatherings of any kind. Performance situations might include times when a person would have to do something in public, such as speak up in class or at a meeting. A person with this condition worries about being embarrassed, or about other people's opinions. People with social phobia usually feel extremely anxious (nervous and worried) about being the focus of attention. They often avoid social and performance situations. This behavior can have a negative effect on the quality of their lives and relationships.

In this study, we want to find out if d-cycloserine can help control social phobia when the drug is added to the standard treatment for this condition. The standard treatment is cognitive-behavior therapy (CBT). CBT is a form of talk therapy involving discussion with a therapist, along with practicing the feelings or events that the person finds frightening.

DETAILED DESCRIPTION:
Inclusion criteria:

1. Age 18 or older
2. Primary diagnosis of SAD
3. Physical examination, electrocardiogram, and laboratory findings without clinically significant abnormalities.
4. Willingness and ability to comply with the requirements of the study protocol.

Diagnostic Exclusion Criteria:

1. A lifetime history of bipolar disorder, schizophrenia, psychosis, delusional disorders or obsessive-compulsive disorder; an eating disorder in the past 6 months; organic brain syndrome, mental retardation or other cognitive dysfunction that could interfere with capacity to engage in therapy; a history of substance or alcohol abuse or dependence (other than nicotine) in the last 6 months or otherwise unable to commit to refraining from alcohol use during the acute period of study participation.
2. Patients with posttraumatic stress disorder within the past 6 months are excluded. Entry of patients with other mood or anxiety disorders will be permitted if the social anxiety disorder is judged to be the predominant disorder, in order to increase accrual of a clinically relevant sample. Patients with significant suicidal ideation (MADRS item 10 score > 3) or who have enacted suicidal behaviors within 6 months prior to intake will be excluded from study participation and referred for appropriate clinical intervention.
3. Patients must be off concurrent psychotropic medication (e.g., antidepressants, anxiolytics, beta blockers) for at least 2 weeks prior to initiation of randomized treatment.
4. Significant personality dysfunction likely to interfere with study participation.
5. Serious medical illness or instability for which hospitalization may be likely within the next year.
6. Patients with a current or past history of seizures
7. Pregnant women, lactating women, and women of childbearing potential who are not using medically accepted forms of contraception (e.g., IUD, oral contraceptives, barrier devices, condoms and foam, or implanted progesterone rods stabilized for at least 3 months).
8. Any concurrent psychotherapy initiated within 3 months of baseline, or ongoing psychotherapy of any duration directed specifically toward treatment of the GSAD is excluded. Prohibited psychotherapy includes CBT or psychodynamic therapy focusing on exploring specific, dynamic causes of the phobic symptomatology and provides management skills. General supportive therapy initiated > 3 months prior is acceptable.
9. Prior non-response to adequately-delivered exposure (i.e., as defined by the patient's report of receiving specific and regular exposure assignments as part of a previous treatment) will exclude participants from the study.
10. Patients with a history of head trauma causing loss of consciousness, seizure or ongoing cognitive impairment.
11. Patients receiving isoniazid.
12. Patients unable to understand study procedures and participate in the informed consent process.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female outpatients > 18 years of age with a primary psychiatric diagnosis (designated by the patient as the most important source of current distress) of generalized social anxiety disorder (GSAD) as defined by DSM-IV criteria.
2. A total score > 60 on the LSAS.
3. Physical examination, electrocardiogram, and laboratory findings without clinically significant abnormalities.
4. Willingness and ability to comply with the requirements of the study protocol.

Exclusion Criteria:

1. A lifetime history of bipolar disorder, schizophrenia, psychosis, delusional disorders or obsessive-compulsive disorder; an eating disorder in the past 6 months; organic brain syndrome, mental retardation or other cognitive dysfunction that could interfere with capacity to engage in therapy; a history of substance or alcohol abuse or dependence (other than nicotine) in the last 6 months or otherwise unable to commit to refraining from alcohol use during the acute period of study participation.
2. Patients with posttraumatic stress disorder within the past 6 months are excluded. Entry of patients with other mood or anxiety disorders will be permitted if the social anxiety disorder is judged to be the predominant disorder, in order to increase accrual of a clinically relevant sample. Patients with significant suicidal ideation (MADRS item 10 score > 3) or who have enacted suicidal behaviors within 6 months prior to intake will be excluded from study participation and referred for appropriate clinical intervention.
3. Patients must be off concurrent psychotropic medication (e.g., antidepressants, anxiolytics, beta blockers) for at least 2 weeks prior to initiation of randomized treatment.
4. Significant personality dysfunction likely to interfere with study participation.
5. Serious medical illness or instability for which hospitalization may be likely within the next year.
6. Patients with a current or past history of seizures
7. Pregnant women, lactating women, and women of childbearing potential who are not using medically accepted forms of contraception (e.g., IUD, oral contraceptives, barrier devices, condoms and foam, or implanted progesterone rods stabilized for at least 3 months).
8. Any concurrent psychotherapy initiated within 3 months of baseline, or ongoing psychotherapy of any duration directed specifically toward treatment of the GSAD is excluded. Prohibited psychotherapy includes CBT or psychodynamic therapy focusing on exploring specific, dynamic causes of the phobic symptomatology and provides management skills. General supportive therapy initiated > 3 months prior is acceptable.
9. Prior non-response to adequately-delivered exposure (i.e., as defined by the patient's report of receiving specific and regular exposure assignments as part of a previous treatment) will exclude participants from the study.
10. Patients with a history of head trauma causing loss of consciousness, seizure or ongoing cognitive impairment.
11. Patients receiving isoniazid.
12. Patients unable to understand study procedures and participate in the informed consent process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2007-03; Primary Completion 2012-03 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Pollack, MD, Principal Investigator — mpollack@partners.org; Stefan Hofmann, Principal Investigator — shofmann@bu.edu
Locations (1):
- Center for Anxiety and Traumatic Stress Disorders, Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Zalta AK, Dowd S, Rosenfield D, Smits JA, Otto MW, Simon NM, Meuret AE, Marques L, Hofmann SG, Pollack MH. Sleep quality predicts treatment outcome in CBT for social anxiety disorder. Depress Anxiety. 2013 Nov;30(11):1114-20. doi: 10.1002/da.22170. Epub 2013 Aug 26. PMID 24038728
- [Derived] Smits JA, Rosenfield D, Otto MW, Marques L, Davis ML, Meuret AE, Simon NM, Pollack MH, Hofmann SG. D-cycloserine enhancement of exposure therapy for social anxiety disorder depends on the success of exposure sessions. J Psychiatr Res. 2013 Oct;47(10):1455-61. doi: 10.1016/j.jpsychires.2013.06.020. Epub 2013 Jul 16. PMID 23870811
- [Derived] Hofmann SG, Smits JA, Rosenfield D, Simon N, Otto MW, Meuret AE, Marques L, Fang A, Tart C, Pollack MH. D-Cycloserine as an augmentation strategy with cognitive-behavioral therapy for social anxiety disorder. Am J Psychiatry. 2013 Jul;170(7):751-8. doi: 10.1176/appi.ajp.2013.12070974. PMID 23599046

RESULTS

PARTICIPANT FLOW:
Groups:
- Cognitive Behavioral Group Therapy + 50mg D-Cycloserine: Participants received Cognitive Behavioral Group Therapy and 50mg D-Cycloserine.
- Cognitive Behavioral Group Therapy + 50mg Placebo: Participants received Cognitive Behavioral Group Therapy and 50mg Placebo.
Period: Overall Study
Arm/Group | Cognitive Behavioral Group Therapy + 50mg D-Cycloserine | Cognitive Behavioral Group Therapy + 50mg Placebo
Started | 87 | 82
Completed | 78 | 69
Not Completed | 9 | 13
Not completed — Lost to Follow-up | 0 | 6
Not completed — Withdrawal by Subject | 8 | 7
Not completed — Hospitalized | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Group Therapy + 50mg D-Cycloserine | Cognitive Behavioral Group Therapy + 50mg Placebo | Total
Number analyzed (Participants) | 87 | 82 | 169
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.6 (10.5) | 30.5 (9.8) | 32.6 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 42 | 73
  Male | 56 | 40 | 96
Region of Enrollment [Number; unit: participants]
  United States | 87 | 82 | 169

OUTCOME MEASURES:

1. Primary Outcome: Liebowitz Social Anxiety Scale (LSAS)
Description: The Liebowitz Social Anxiety Scale (LSAS) is a 24-item measure designed to assess both fear and avoidance of social and performance situations occurring in the last week. Each item is rated from 0-3 for both fear and avoidance with a possible score of 144; 55-65 Moderate social phobia, 65-80 Marked social phobia, 80-95 Severe social phobia, and Greater than 95 - Very severe social phobia. Remission was defined as a score of < 30 on the Liebowitz Social Anxiety Scale
Time Frame: Week 13
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Cognitive Behavioral Group Therapy + 50mg D-Cycloserine | Cognitive Behavioral Group Therapy + 50mg Placebo
Number analyzed (Participants) | 87 | 82
units on a scale | 39.19 [34.79 to 43.59] | 42.44 [37.94 to 47.03]

2. Primary Outcome: CGI - Clinical Global Impression of Improvement
Description: The Clinician Global Impression-Improvement Scale (CGI-I) is a clinician-rated instrument used to assess global severity of symptoms. The CGI-I ranges from 1 ("very much improved") to 7 ("very much worse"). Response and remission was defined as an improvement score of 1 ("very much improved") or 2 ("much improved") on the CGI-I.
Time Frame: Week 13
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Cognitive Behavioral Group Therapy + 50mg D-Cycloserine | Cognitive Behavioral Group Therapy + 50mg Placebo
Number analyzed (Participants) | 87 | 82
units on a scale | 2.68 [2.38 to 2.98] | 2.95 [2.64 to 3.27]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 6 weeks.
Description: Patients were asked about the occurrence of adverse events during each visit. These will be recorded by the clinician on the Adverse Events form and rated as mild, moderate or severe.
Groups:
- Cognitive Behavioral Therapy + DCS: Participants received Cognitive Behavioral Group Therapy and 50mg D-Cycloserine.
- Cognitive Behavioral Therapy + Placebo: Participants received Cognitive Behavioral Group Therapy and Placebo.
Arm/Group | Cognitive Behavioral Therapy + DCS | Cognitive Behavioral Therapy + Placebo
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/82
Other Adverse Events (participants affected / at risk) | 26/87 | 19/82
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cognitive Behavioral Therapy + DCS (N=87) | Cognitive Behavioral Therapy + Placebo (N=82)
General (General disorders) | 7 | 4
Neurological (General disorders) | 6 | 4
GI (General disorders) | 5 | 4
Cognitive/Emotional (General disorders) | 3 | 1
Genitourinary (General disorders) | 0 | 1
Other (General disorders) | 6 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No